CLINICAL TRIAL: NCT02791399
Title: A Patient-Centered Intervention to Improve Opioid Safety
Acronym: ISOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 14-020; 9024 (Other Grant/Funding Number: VA - Health Services R&D)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Opioid Safety; Prescription Opioid Misuse; Chronic Pain
Keywords: opioid safety; opioid misuse; opioid abuse; patient-centered; opioid; opiate; chronic pain; primary care; Veteran; clinical care
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Treatment as usual
- ISOP Intervention (Experimental): Primary care providers and PACT nurses will participate in the same workshop as those randomized to the control condition (or academic detailing for those unable to attend the workshop). Clinicians randomized to the intervention will additionally collaborate with a nurse care manager (NCM) who will maintain a registry of enrolled patients, track UDT administrations and results, query prescription drug monitoring databases, monitor other evidence of potential problems, and collaborate with expert consultants to provide decision support when patients have evidence of prescription opioid misuse or abuse. The NCM will also meet with patients to discuss methods to reduce opioid adverse effects, prevent misuse, and provide rationale for prescription opioid adherence monitoring.
  Interventions: Behavioral: ISOP Intervention with the Nurse Care Manager

INTERVENTIONS:
Behavioral: ISOP Intervention with the Nurse Care Manager — A Nurse Care Manager (NCM) will maintain a registry of enrolled patients, track opioid medication-related events from the medical record, and provide decision support to Primary Care Providers for issues related to prescription opioid safety. The NCM will also meet individually with enrolled participants in the intervention group to discuss strategies for preventing/reducing opioid side effects, preventing diversion, and providing rationale for screening for prescription opioid misuse.
  Arms: ISOP Intervention

SUMMARY:
This is a randomized controlled trial of a multifaceted intervention designed to improve the safety of opioid prescribing. The specific aims of this study are to: (a) evaluate whether a multifaceted intervention (Improving the Safety of Opioid Prescribing; ISOP) enhances opioid safety, (b) assess whether participation in ISOP impacts the clinician-patient relationship, and (c) explore to what extent ISOP is associated with changes in pain and pain-related function.

DETAILED DESCRIPTION:
The investigators will randomize primary care providers (PCPs) at the VA Portland Health Care System to either ISOP or the control condition; patients will be nested by clinician status. All PCPs who enroll will participate in either a two-hour educational workshop or the two-hour educational workshop + nurse care manager (NCM). The NCM will maintain a registry of enrolled patients, track opioid medication-related events from the medical record, and provide decision support to PCPs for issues related to prescription opioid safety. The NCM will also meet individually with enrolled participants to discuss strategies for preventing/reducing opioid side effects, preventing diversion, and providing rationale for screening for prescription opioid misuse. The investigators will recruit patients who are already prescribed chronic opioid therapy for chronic non-cancer pain. Participants will be enrolled for one year. Outcomes will be measured at baseline, and 6 and 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in primary care at the VA Portland Health Care System
* Receiving long-term opioid therapy (for at least 3 months) for chronic pain unrelated to a life-limiting disease
* Able to read and write in English

Exclusion Criteria:

* Age younger than 18 years old
* On opioid therapy for palliative or end-of-life care
* Current enrollment in an opioid substitution program
* Lack of access to a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J. Morasco, PhD MA, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maloy PE, Iacocca MO, Morasco BJ. CE: Implementing Guidelines for Treating Chronic Pain with Prescription Opioids. Am J Nurs. 2019 Nov;119(11):22-29. doi: 10.1097/01.NAJ.0000605344.99391.78. PMID 31651495
- [Result] Morasco BJ, Adams MH, Maloy PE, Hooker ER, Iacocca MO, Krebs EE, Carr TP, Lovejoy TI, Saha S, Dobscha SK. Research methods and baseline findings of the improving the safety of opioid therapy (ISOT) cluster-randomized trial. Contemp Clin Trials. 2020 Mar;90:105957. doi: 10.1016/j.cct.2020.105957. Epub 2020 Feb 13. PMID 32061968
- [Result] Morasco BJ, Iacocca MO, Lovejoy TI, Dobscha SK, Deyo RA, Cavese JA, Hyde S, Yarborough BJH. Utility of the Pain Medication Questionnaire to predict aberrant urine drug tests: Results from a longitudinal cohort study. Psychol Serv. 2021 Aug;18(3):319-327. doi: 10.1037/ser0000471. Epub 2020 Jul 16. PMID 32673038
- [Result] Wilson AC, Morasco BJ, Holley AL, Feldstein Ewing SW. Patterns of opioid use in adolescents receiving prescriptions: The role of psychological and pain factors. Am Psychol. 2020 Sep;75(6):748-760. doi: 10.1037/amp0000697. PMID 32915020
- [Result] Bryson WC, Morasco BJ, Cotton BP, Thielke SM. Cannabis Use and Nonfatal Opioid Overdose among Patients Enrolled in Methadone Maintenance Treatment. Subst Use Misuse. 2021;56(5):697-703. doi: 10.1080/10826084.2021.1892137. Epub 2021 Mar 22. PMID 33749499
- [Result] Magaletta PR, Morasco BJ. Perspectives on opioid misuse from public service psychology: An introduction. Psychol Serv. 2021 Aug;18(3):285-286. doi: 10.1037/ser0000485. PMID 34370491
- [Result] Borsari B, Li Y, Tighe J, Manuel JK, Gokbayrak NS, Delucchi K, Morasco BJ, Abadjian L, Cohen BE, Baxley C, Seal KH. A pilot trial of collaborative care with motivational interviewing to reduce opioid risk and improve chronic pain management. Addiction. 2021 Sep;116(9):2387-2397. doi: 10.1111/add.15401. Epub 2021 Jan 27. PMID 33405304
- [Result] Morasco BJ, Smith N, Dobscha SK, Deyo RA, Hyde S, Yarborough BJ. Prospective Investigation of Factors Associated with Prescription Opioid Dose Escalation among Patients in Integrated Health Systems. J Gen Intern Med. 2020 Dec;35(Suppl 3):895-902. doi: 10.1007/s11606-020-06250-x. Epub 2020 Nov 3. PMID 33145684
- [Result] Morasco BJ, Adams MH, Hooker ER, Maloy PE, Krebs EE, Lovejoy TI, Saha S, Dobscha SK. A Cluster-Randomized Clinical Trial to Decrease Prescription Opioid Misuse: Improving the Safety of Opioid Therapy (ISOT). J Gen Intern Med. 2022 Nov;37(15):3805-3813. doi: 10.1007/s11606-022-07476-7. Epub 2022 Mar 16. PMID 35296983

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | ISOP Intervention
Started | 136 | 150
Completed | 123 | 135
Not Completed | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | ISOP Intervention | Total
Number analyzed (Participants) | 136 | 150 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.8) | 61.2 (10.9) | 60.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 115 | 135 | 250
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 108 | 123 | 231
  African-American | 6 | 5 | 11
  Native American or Alaska Native | 10 | 15 | 25
  Asian or Pacific Islander | 1 | 2 | 3
  Other | 11 | 5 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 136 | 150 | 286
Marital status [Count of Participants; unit: Participants]
  Single or never married | 8 | 10 | 18
  Divorced or separated | 42 | 41 | 83
  Married or living with partner | 80 | 89 | 169
  Widowed | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Current Opioid Misuse Measure (COMM)
Description: The Current Opioid Misuse Measure (COMM) is an assessment of self-reported risk of prescription opioid misuse. There are 17 items, each rated on a scale of 0 (never) to 4 (very often). Total scores range from 0 - 68, with higher scores indicating a greater risk of prescription opioid misuse.
Time Frame: Data collected at baseline, 6 months, and 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | ISOP Intervention
Number analyzed (Participants) | 123 | 135
score on a scale
  Baseline | 11.3 (8.0) | 11.9 (6.8)
  6 month follow-up | 9.4 (6.4) | 9.5 (6.7)
  12 month follow-up | 9.3 (6.5) | 8.6 (5.7)
Statistical Analysis 1: Comparison: Control vs ISOP Intervention; Test type: Equivalence — Our analysis examined the estimated averages for each group at each time point after accounting for covariates; p < 0.05, Mixed Models Analysis; Models controlled for age, gender, depression severity, pain intensity, clinician type, and proportion of clinician panel prescribed opioids; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-2.45 to 0.20]

2. Primary Outcome: Urine Drug Test
Description: Participants will complete urine drug tests (UDTs) to evaluate for presence of substances. UDTs will evaluate for cannabis, cocaine, amphetamines, benzodiazepines, barbiturates, opioids, and opiates. Study results are dichotomous.
Time Frame: Data collected at baseline, 6 months, and 12 months
Population: Smaller n due to missing values.
Measure: Number; unit: percentage of aberrant UDT results
Arm/Group | Control | ISOP Intervention
Number analyzed (Participants) | 125 | 138
percentage of aberrant UDT results
  Baseline | 12.8 | 10.9
  6 months | 7.0 | 14.0
  12 months | 16.2 | 10.2
Statistical Analysis 1: Comparison: Control vs ISOP Intervention; Test type: Equivalence — Our analysis examined the estimated probabilities for each group at each time point after accounting for covariates; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.15 to 0.06]

3. Secondary Outcome: Chronic Pain Grade
Description: The Chronic Pain Grade is a 7-item self-report measure that provides global scores of pain intensity and function. Scores for each subscale range from 0 - 100. Higher scores indicate more severe pain or more impairment in function. Pain intensity and function were tested in a non-inferiority analysis.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | ISOP Intervention
Number analyzed (Participants) | 136 | 150
score on a scale | 65.8 (15.5) | 67.0 (14.5)
Statistical Analysis 1: Comparison: Control vs ISOP Intervention; Test type: Non-Inferiority — Pain intensity and pain-related function were tested in non-inferiority analyses, as we hypothesized that the ISOT intervention would not negatively impact pain or function. One-half SD difference in change was considered the appropriate non-inferiority limit; Non-inferiority analysis = 1.60

4. Other Pre Specified Outcome: Trust in Physician Scale
Description: The Trust in Physician Scale is an 11-item self-report measure. Scores range from 0 - 100, with higher scores indicating greater interpersonal trust between patients and their clinician
Time Frame: Data collected at baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | ISOP Intervention
Number analyzed (Participants) | 136 | 150
score on a scale
  Baseline | 66.3 (18.6) | 66.8 (20.2)
  6 months | 68.0 (18.6) | 66.5 (21.9)
  12 months | 68.1 (18.0) | 65.9 (21.2)
Statistical Analysis 1: Comparison: Control vs ISOP Intervention; Test type: Equivalence — This analysis is comparing estimated averages and probabilities for each group at each time point after accounting for covariates; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-5.83 to 1.85]

5. Other Pre Specified Outcome: Participatory Decision Making Style
Description: The Participatory Decision Making Style is a 4-item self-report measures. Scores range from 0 - 100, where higher scores indicate greater patient involvement in medical decision making.
Time Frame: Data collected at baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | ISOP Intervention
Number analyzed (Participants) | 136 | 150
score on a scale
  Baseline | 50.3 (32.4) | 50.4 (35.7)
  6 months | 57.6 (31.9) | 51.9 (36.9)
  12 months | 54.3 (33.5) | 55.1 (34.9)
Statistical Analysis 1: Comparison: Control vs ISOP Intervention; Test type: Equivalence — Our analysis examined the estimated averages for each group at each time point after accounting for covariates; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-6.73 to 8.80]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | ISOP Intervention
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/150
Other Adverse Events (participants affected / at risk) | 0/136 | 0/150

LIMITATIONS AND CAVEATS:
Had planned to study changes in rates of substance use disorders (measured with the SCID). However, due to low enrollment of participants with SUD, groups comparisons on changes in SUD rates were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT02791399/Prot_SAP_000.pdf